CLINICAL TRIAL: NCT05379881
Title: An Online Wellness Intervention: Investigating the Efficacy of the Common Elements Toolbox
Brief Title: Efficacy of COMET on Prolific Participants
Acronym: COMET-Prol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Lorenzo Lorenzo-Luaces, Assistant Professor Pyschological and Brain Sciences, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12290
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Depression; Anxiety; Emotion Regulation
MeSH Terms: conditions — Depression; Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waiting list control (WLC) (No Intervention): Participants who are assigned to the control condition will complete the baseline questionnaires and assessments at weeks 2, 4, and 8. After the last assessment, they will be given access to COMET.
- Common Elements Toolbox (COMET) (Experimental): COMET consists of the following modules: cognitive restructuring (labeled "flexible thinking"), behavioral activation (labeled "positive activities"), gratitude, and self-compassion. Participants complete these COMET modules by themselves. The format is reading psychoeducational along with completing specific activities.
  Interventions: Behavioral: Common Elements Toolbox (COMET)

INTERVENTIONS:
Behavioral: Common Elements Toolbox (COMET) — COMET is an unguided single-session intervention (SSI) combining elements of cognitive-behavioral therapy (CBT) and positive psychology.
  Other Names: single session intervention; unguided self-help; internet-based CBT
  Arms: Common Elements Toolbox (COMET)

SUMMARY:
In this study, the investigators will test the effectiveness of a digital, single-session mental health intervention. There will be two conditions: the COMET intervention and the control group. The program, COMET (Common Elements Toolbox), will include a variety of modules which will focus on cognitive restructuring, gratitude, behavioral activation, and self-compassion. A similar intervention has previously been tested with Indian adolescents and adapted for US graduate students.

DETAILED DESCRIPTION:
Participants who follow the study link in Prolific will immediately be taken to the Informed Consent Statement (ICS), which will include a description of the study, risks and benefits, payment, and confidentiality. After reading the ICS, participants will confirm their consent by clicking "I consent to participate in this study." They will then be taken to the welcome page for the study and confirm that they will provide their best answers. Once participants have confirmed their consent, they will be taken to the rest of the survey.

All participants will fill out a series of questionnaires including: the Generalized Anxiety Disorder 7-item (GAD-7), Patient Health Questionnaire 8-item (PHQ-8), WHO-5 Wellbeing Index (WHO-5), 3 questions from the Insomnia Severity Index (ISI), Emotion Regulation Questionnaire (ERQ), Ten-Item Personality Inventory (TIPI), Adverse Childhood Experiences Scale (ACES), Work and Social Adjustment Scale (WSAS), 4 mechanisms questions, 3 items from the Secondary Control Scale (SCS), Module preferences and the System Usability Scale (SUS). After completing these questionnaires participants will be randomized to either the COMET intervention condition (who receive the intervention immediately) or the control condition (who will receive the intervention after 8 weeks). they will be randomized to one of two conditions: COMET (will receive the COMET intervention immediately) or a waitlist control (will receive the COMET intervention in 8 weeks). This randomization will be completed via the Qualtrics randomizer function - which randomly and evenly assigns participants to the two conditions.

Participants who are assigned to the COMET condition will then be taken to the intervention introduction. They will then receive the following modules: cognitive restructuring (labeled "flexible thinking"), behavioral activation (labeled "positive activities"), gratitude, and self-compassion. In the flexible thinking module, participants will learn to identify and reframe negative beliefs. They will first read about a hypothetical character who is adjusting to changes in their routine. Then, using the character's story as an example, they will try to identify negative beliefs that the character may be experiencing and ways the character could reframe the belief. Then, they will apply this technique to a situation in their own life. In the positive activities module, participants will identify and reflect on activities that are important to them. They will list activities they find enjoyable and meaningful. Then, they will reflect on why these activities matter to them and schedule in time to perform these activities in the weeks ahead. In the gratitude module, participants will be asked to reflect and write about 3 things they are grateful about. They will then be asked to think and write about things they notice around them that they enjoy and are grateful for. In the self-compassion module, participants will be asked to write a self-compassion letter to themselves, expressing compassion towards themselves just as they would towards a friend or family member. They will also be requested to create a few sentences that they would like to hear when feeling self-critical.

After completing the COMET intervention, participants will complete the post-intervention questions. A mental wellbeing resource list will be provided at the end of the session.

Participants who are assigned to the control condition will complete a separate series of questionnaires: hypothetical questions about emotional experiences using questions from the GAD-7 (Hypothetical Questions - GAD-7) and hypothetical questions about emotional experiences using questions from the PHQ-9 (Hypothetical Questions - PHQ-9).

After completing the COMET intervention or completing the control questions, all participants will fill out demographic information including age, sex assigned at birth, gender, race/ethnicity, sexual orientation, relationship status, how often they attend religious services, education level, annual income, employment status, if they have ever taken anti-depressants or other psychiatric medication, how many people they can rely on for social support, physical health, how often they drink alcohol, and how old they were when they first struggled with depression, anxiety, or stress.

All participants in both conditions will be invited via Prolific to continue to complete measures at follow-up time points of 2 weeks, 4 weeks, and 8 weeks post-baseline (approx. 10-15 minutes each). In the informed consent statement, participants will be informed that there are follow-up assessments that they can receive additional compensation for. There will also be reminders at the end of the baseline assessment reminding them to watch for the follow ups. They will not be notified of these follow-up assessments, but will be able to see the follow-up assessments posted on Prolific. During these follow-ups all participants (e.g., those in both the intervention and control conditions) will complete the following questionnaires: GAD-7, PHQ-8, WHO-5, ISI, ERQ, WSAS, and SCS.

After completing the follow-up measure at 8 weeks, enrollment in the study will end. At this point, participants in the control condition will receive the intervention modules. Their use of the COMET intervention is entirely optional and will not be recorded by the research team. They will not fill out any follow up measures after completing or not completing the COMET intervention.

Below is a complete schedule for participants in the study, separated by condition (e.g., COMET vs control).

COMET INTERVENTION

Baseline:

Measures/questionnaires (pre-intervention): Informed consent statement --> Intro Text --> Generalized Anxiety Disorder 7-item (GAD-7), Patient Health Questionnaire 8-item (PHQ-8), WHO-5 Wellbeing Index (WHO-5), 3 questions from the Insomnia Severity Index (ISI), Emotion Regulation Questionnaire (ERQ), Ten-Item Personality Inventory (TIPI), Adverse Childhood Experiences Scale (ACES), Work and Social Adjustment Scale (WSAS), 4 mechanisms questions, 3 items from the Secondary Control Scale (SCS), Module preferences and the System Usability Scale (SUS).

Intervention: After filling out these questionnaires, they will proceed to the COMET intervention content, which consists of the intervention introduction and 4 modules - cognitive restructuring (labeled "flexible thinking"), behavioral activation (labeled "positive activities"), gratitude, and self-compassion.

Measures/questionnaires (post-intervention): Post Intervention Questions, demographic information.

Time to complete: approximately 60-80 minutes.

2-week follow up: Measures/questionnaires: GAD-7, PHQ-8, WHO-5, ISI, ERQ, WSAS, and SCS. Time to complete: approximately 10-15 minutes.

4-week follow up: Measures/questionnaires: GAD-7, PHQ-8, WHO-5, ISI, ERQ, WSAS, and SCS. Time to complete: approximately 10-15 minutes.

8-week follow up: Measures/questionnaires: GAD-7, PHQ-8, WHO-5, ISI, ERQ, WSAS, and SCS. Time to complete: approximately 10-15 minutes.

CONTROL CONDITION

Baseline:

Measures/questionnaires: Informed consent statement --> Intro Text --> Generalized Anxiety Disorder 7-item (GAD-7), Patient Health Questionnaire 8-item (PHQ-8), WHO-5 Wellbeing Index (WHO-5), 3 questions from the Insomnia Severity Index (ISI), Emotion Regulation Questionnaire (ERQ), Ten-Item Personality Inventory (TIPI), Adverse Childhood Experiences Scale (ACES), Work and Social Adjustment Scale (WSAS), 4 mechanisms questions, 3 items from the Secondary Control Scale (SCS), Module preferences and the System Usability Scale (SUS); hypothetical questions about emotional experiences using questions from the GAD-7 (Hypothetical Questions - GAD-7); hypothetical questions about emotional experiences using questions from the PHQ-9 (Hypothetical Questions - PHQ-9); demographic information.

Time to complete: approximately 15-20 minutes.

2-week follow up: GAD-7, PHQ-8, WHO-5, ISI, ERQ, WSAS, and SCS. Time to complete: approximately 10-15 minutes.

4-week follow up: GAD-7, PHQ-8, WHO-5, ISI, ERQ, WSAS, and SCS. Time to complete: approximately 10-15 minutes.

8-week follow up: GAD-7, PHQ-8, WHO-5, ISI, ERQ, WSAS, and SCS. Time to complete: approximately 10-15 minutes.

After completing the 8-week follow up, participants in the control condition will be sent the COMET intervention modules. Whether they complete the intervention or not is entirely up to them and it will not be tracked by the research team.

ELIGIBILITY:
Inclusion Criteria:

* A positive response (i.e., "yes") to the question: "Do you have or have you had a diagnosed, ongoing mental health/illness/condition?"

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2022-09-03 (Actual)

PRIMARY OUTCOMES:
2-week change in the Patient Health Questionnaire | 2 weeks
  Changes in PHQ8 from baseline to Week 2. The PHQ8 is a measure of depression and the measure is scored on a scale of 0 - 24 where higher scores indicate higher depression (i.e., are negative). Thus, lower scores relative to baseline indicate more positive outcomes.
2-week change in the Generalized Anxiety Disorder 7 scale (GAD7) | 2 weeks
  Changes in GAD7 from baseline to Week 2. The GAD7 is a measure of anxiety and the measure is scored on a scale of 0 - 21 where higher scores indicate higher anxiety (i.e., are negative). Thus, lower scores relative to baseline indicate more positive outcomes.
8-week change in the Patient Health Questionnaire | 8 weeks
  Changes in PHQ8 from baseline to Week 8. The PHQ8 is a measure of depression and the measure is scored on a scale of 0 - 24 where higher scores indicate higher depression (i.e., are negative). Thus, lower scores relative to baseline indicate more positive outcomes.
8-week change in the Generalized Anxiety Disorder 7 scale (GAD7) 8-week change in the Generalized Anxiety Disorder 7 scale (GAD7) | 8 weeks
  Changes in GAD7 from baseline to Week 2. The GAD7 is a measure of anxiety and the measure is scored on a scale of 0 - 21 where higher scores indicate higher anxiety (i.e., are negative). Thus, lower scores relative to baseline indicate more positive outcomes.

SECONDARY OUTCOMES:
8-week change in the World Health Organization Well-being Index 5 (WHO5) | 8 weeks
  Changes in WHO-5 from baseline to 8 weeks after the termination of the study. The WHO-5 is a measure of well-being and the measure is scored on a scale of 0 - 100 where higher scores indicate higher satisfaction with life (i.e., are positive). Thus, higher scores relative to baseline indicate more positive outcomes.
8-week change in the Work and Social Adjustment Scale (WSAS) | 8 weeks
  Changes in WSAS from baseline to Week 8. The WSAS is a measure of impairment in functioning and the measure is scored on a scale of 0 - 40 where higher scores indicate great dysfunction (i.e., are negative). Thus, lower scores relative to baseline indicate more positive outcomes.
8-week change in Emotion Regulation Scale (ERQ) - Reappraisal subscale | 8 weeks
  Changes in the ERQ Reappraisal subscale from baseline to Week 8. The Reappraisal scale is a measure of regulating emotions by engaging in reappraisal (i.e., changing the one one thinks about an emotion evoking stimuli), widely considered an adaptive strategy. The measured is scored on a 1-7 scale where higher scores indicate greater use of adaptive emotion regulation strategies (i.e., positive). Thus, higher scores relative to baseline indicate more positive outcomes.
8-week change in the Emotion Regulation Scale (ERQ) - Suppression subscale | 8 weeks
  Changes in the ERQ Suppression Scale from baseline to Week 8. The ERQ Suppression scale is a measure of regulating emotions by engaging in suppression (i.e., trying not to think or feel), which is considered a maladaptive emotion regulation strategy. The measure is scored on a scale of 1 - 7 where higher scores indicate higher use of suppression (i.e., negative). Thus, lower scores relative to baseline indicate more positive outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorenzo-Luaces L, Howard J. Efficacy of an Unguided, Digital Single-Session Intervention for Internalizing Symptoms in Web-Based Workers: Randomized Controlled Trial. J Med Internet Res. 2023 Jul 7;25:e45411. doi: 10.2196/45411. PMID 37418303